CLINICAL TRIAL: NCT06996366
Title: Reducing Racial and Ethnic Disparities in Medicare Annual Wellness Visit Uptake
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, David Liss, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00219825; R21AG081895-01A1 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Annual Wellness Visit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early outreach (Experimental): Patients assigned to early outreach will receive mailed letter and telephone outreach encouraging them to schedule an Annual Wellness Visit with a primary care clinician. Social determinants of health screening and resource provision if applicable will be included in telephone outreach by health navigator.
  Interventions: Other: Outreach to encourage Annual Wellness Visit completion
- Delayed outreach (Other): Patients assigned to delayed outreach will receive no outreach for 6 months after study start and then will receive the same outreach intervention as early outreach arm.
  Interventions: Other: Outreach to encourage Annual Wellness Visit completion

INTERVENTIONS:
Other: Outreach to encourage Annual Wellness Visit completion — Mailed and telephone outreach to patient.

SUMMARY:
The goal of this randomized pilot study is to learn the impact of a primary care outreach intervention on the proportion of patients with Medicare insurance who are up-to-date on Medicare Annual Wellness Visit completion. At two clinics, researchers will randomize clinicians (and their associated, eligible patients) to early or delayed outreach.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 in-person primary care visit during 18-month lookback period AND
* Medicare or Medicare Advantage insurance AND
* ≥1 risk factor shown to be associated with being overdue for Medicare Annual Wellness Visits (identified in preparatory analysis prior to pilot trial): Black/African American race or Latino/Hispanic ethnicity OR Not up-to-date for social needs screening OR Positive social need in past 18 months OR Medicaid insurance OR No use of scheduling features within patient portal in past 18 months
* Preferred language English AND
* Attributed primary care clinic is 1 of the participating clinics in the pilot trial AND
* No AWV completion (CPT G0402, G0438, G0439, G0468) during 10-month lookback period AND
* No appointment scheduled for upcoming AWV

Exclusion Criteria:

* Patients will be excluded if they are receiving palliative care or if their clinician feels that outreach for preventive care is inappropriate.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 174 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Completion of Annual Wellness Visit | 6 months
  Binary (0/1) patient-level measure, based on presence of any CPT (Current Procedural Terminology) codes for Medicare preventive visits during follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No